CLINICAL TRIAL: NCT02997553
Title: Reliability of Indocyanine Green Use in Sentinel Lymph Node Identification in Cancer Surgery
Brief Title: Fluorescence for Sentinel Lymph Node Identification in Cancer Surgery
Acronym: GASVERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00799-42
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Breast Carcinoma; Head and Neck Cancer; Melanoma (Skin); Squamous Cell Carcinoma, Skin; Cervix Cancer; Endometrium Cancer; Ovary Cancer; Vulva Cancer; Anus Cancer; Rectum Cancer
Keywords: Indocyanine green (ICG); Sentinel lymph node biopsy; Technetium99; Tumors; Optonuclear probe; Surgery
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Melanoma; Carcinoma, Squamous Cell; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Rectal Neoplasms; Neoplasms | interventions — Indocyanine Green; Infracyanine green; Technetium-99; nanocis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sentinel lymph node detection (Experimental): Each patient receive both injections of Technetium99 (standard care) and indocyanine green.
  The detection of sentinel lymph node will be conducted by an optonuclear probe able to detect the radioactive and the fluorescence signal during surgery.
  Interventions: Drug: Indocyanine green; Drug: Technetium99; Device: Optonuclear probe; Device: Quest Camera

INTERVENTIONS:
Drug: Indocyanine green — Each patient receive injection of indocyanine green just before surgery Specify total dose : 2.5 mg/ml (Intravenous use)
  Other Names: Infracyanine
Drug: Technetium99 — Each patient receives injection of Technetium 99 ( injected in subcutaneously) before surgery.
  Lymphoscintigraphy is performed to identify the sentinel node
  Other Names: NANOCIS
Device: Optonuclear probe — The detection of sentinel lymph node will be conducted by an optonuclear probe able to detect the radioactive and the fluorescence signal during surgery.
Device: Quest Camera — The detection of sentinel lymph node will be conducted by a camera able to determine imagery of fluorescence during surgery.

SUMMARY:
This is a single-center prospective clinical trial to evaluate non-inferiority of indocyanine green guided sentinel lymph node biopsy compared with the gold standard Technecium99 guided sentinel lymph node biopsy in patients with cancers and subjected to surgery.

The diagnostic performance and the tolerance of indocyanine green (ICG) to the radio-isotope (Techniciun99) in the detection of sentinel lymph nodes will be assess using an "Optonuclear" probe (EURORAD S.A.) and QUEST camera

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* cancer histologically proved
* patient eligible for sentinel node detection
* contraceptive methods for men and women of childbearing age
* signed informed consent form
* patient affiliated to the social security system

Exclusion Criteria:

* neoadjuvant chemotherapy or hormone therapy
* adenopathy (s) clinically suspicious or positively cytopenic
* women who are pregnant or breast-feeding
* associated pathology that may prevent patient of receive indocyanine green
* ongoing participation in another clinical trial with an investigational drug
* patients deprived of liberty or under supervision
* impossibility to undergo medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of indocyanine green guided sentinel lymph node biopsy | 1 day
  The detection rate is defined by the number of patient who at least one sentinel node detected by fluorescence or isotope intra operatively.
  Per-operative detection is defined by the identification of at least one sentinel lymph node in the lymphatic drainage area.

SECONDARY OUTCOMES:
Total number of sentinel lymph node detected | 1 day
  The total number of sentinel node detected will be assess by the two techniques
Number of false negative result | 1 day
  False negative result is defined by number of patients with at least one hot metastatic sentinel lymph node without fluorescent metastatic sentinel lymph node
Allergic reactions | 8 days
  Percentage of patients with allergic reactions
Evaluation of pain | 1 day
  Pain will be assessed by a numerical scale from 0 (no pain) to 10 (maximum pain)
fluorescence imaging | 1 day
  The total number of sentinel node detected by fluorescence imaging

CONTACTS AND LOCATIONS:
Overall Officials: MARCHAL FREDERIC, MD, PU-PH, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No